CLINICAL TRIAL: NCT01493388
Title: Observational, Cross-sectional and Retrospective Study on Diabetes Mellitus Type 1 in Tunisian Children and Adolescents Under 15 Years
Brief Title: To Estimate the Percentage of Children and Adolescents in Tunisia With Acceptably Controlled Diabetes Mellitus Type 1
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: INS-3914; U1111-1124-9862 (Other: WHO)
Record Dates: First submitted 2011-12-14; First posted 2011-12-16 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: insulin

INTERVENTIONS:
Drug: insulin — Patients will be treated according to routine clinical practice at the discretion of the treating physician.

SUMMARY:
This study is conducted in Africa. The aim of this study is to estimate the percentage of children and adolescents below or equal to 15 years in Tunisia with acceptably controlled diabetes mellitus type 1.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained before any study-related activities. (Study-related activities are any procedure related to recording of data according to the protocol).
* Child or adolescent below or equal to 15 years with diabetes mellitus type 1
* Who has been undergoing treatment for diabetes for at least 6 months

Exclusion Criteria:

* Previous participation in this study.
* Current participation to a clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be treated according to routine clinical practice at the discretion of the treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 402 (Actual)
Dates: Start 2012-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Percentage of children below 6 years with HbA1c less than 8.5% | one assessment during a 5 month period is made, by review of the patient's medical records and/or interview (only 1)
Percentage of children between 6-12 years with HbA1c less than 8% | one assessment during a 5 month period is made, by review of the patient's medical records and/or interview (only 1)
Percentage of adolescents between 13 and 15 years with HbA1c less than 7.5% | one assessment during a 5 month period is made, by review of the patient's medical records and/or interview (only 1)

SECONDARY OUTCOMES:
Fasting plasma glucose (FPG) level | one assessment during a 5 month period is made, by review of the patient's medical records and/or interview (only 1)
Blood pressure level in children 12 years or older | one assessment during a 5 month period is made, by review of the patient's medical records and/or interview (only 1)
Total cholesterol and LDL-cholesterol levels in children 12 years or older | one assessment during a 5 month period is made, by review of the patient's medical records and/or interview (only 1)
Percentage of children with evaluation of thyroid function within the last 2 years | one assessment during a 5 month period is made, by review of the patient's medical records and/or interview (only 1)
Percentage of children with nephropathy | one assessment during a 5 month period is made, by review of the patient's medical records and/or interview (only 1)
Percentage of children with microalbuminuria | one assessment during a 5 month period is made, by review of the patient's medical records and/or interview (only 1)
Percentage of children with hypoglycemia event having led to hospitalization | one assessment during a 5 month period is made, by review of the patient's medical records and/or interview (only 1)
Percentage of children with self-monitoring of blood-glucose | one assessment during a 5 month period is made, by review of the patient's medical records and/or interview (only 1)
Percentage of parents and children having received at least one training and topic of the received training | one assessment during a 5 month period is made, by review of the patient's medical records and/or interview (only 1)
Type and dose of insulin treatment | one assessment during a 5 month period is made, by review of the patient's medical records and/or interview (only 1)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tunisia, Tunisia

REFERENCES:
- [Result] Hachicha M, Kamoun T, Briki S, Ouamara N. Étude observationnelle sur le diabète de type 1 chez les enfants et les adolescents de moins de 15 ans. La Revue Maghrebine d'Endocrinologie - Diabète et Reproduction; 19 (4): 144-149
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com